CLINICAL TRIAL: NCT00786318
Title: Prospective Double Blind Randomized Trial of Intramuscular Ziprasidone Compared With Standard Antipsychotic Therapy For The Treatment Of The Acutely Agitated Patient In The Emergency Department
Brief Title: Ziprasidone vs Standard Therapy for Agitated Patients in the ED
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor terminated
Sponsor: George Washington University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Jeremy Brown, Dept of Emergency Medicine, The George Washington University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 010411 (completed)
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Psychosis; Agitation; Delirium
Keywords: Psychosis; Agitation; Delirium
MeSH Terms: conditions — Psychotic Disorders; Psychomotor Agitation; Delirium | interventions — ziprasidone; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ziprasidone (Experimental)
  Interventions: Drug: ziprasidone
- Standard therapy (Active Comparator)
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: ziprasidone — ziprasidone 20mg IM
  Arms: ziprasidone
Drug: Standard therapy — Haldol 5mg/ Ativan 2mg IM
  Arms: Standard therapy

SUMMARY:
The primary objective is to determine if ziprasidone is superior to standard therapies in the emergency department treatment of the acutely agitated patient. The primary outcome will be the length of time taken until the patient is ready to be evaluated by the psychiatric service, or until a disposition is made.

ELIGIBILITY:
Inclusion Criteria:

* Acutely agitated
* Requires chemical sedation

Exclusion Criteria:

* Physician preference for a specific chemical sedative
* Known allergy to any study medications

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
length of time from triage until patient is either ready to be seen by psychiatry or is ready to have a disposition made | During ED stay

SECONDARY OUTCOMES:
Length of time taken to sedate patient | Ed visit
Total time spent in restraints | ED visit
Cost effectiveness of the therapy | ED visit

CONTACTS AND LOCATIONS:
Locations (1):
- The George Washington University Medical Center, Dept of Emergency Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Brown J. The spectrum of informed consent in emergency psychiatric research. Ann Emerg Med. 2006 Jan;47(1):68-74. doi: 10.1016/j.annemergmed.2005.08.025. Epub 2005 Nov 17. PMID 16387220